CLINICAL TRIAL: NCT04388930
Title: Longitudinal Characterisation of the Host Microbiota After Kidney Donation and Transplantation
Brief Title: The Microbiota in Kidney Donation and Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: 125570
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Kidney Diseases; Kidney Transplant Failure and Rejection; Urinary Tract Infections
MeSH Terms: conditions — Kidney Diseases; Rejection, Psychology; Urinary Tract Infections | interventions — Urination; Postoperative Period

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and faecal samples will be characterised and compared between pre- and post-surgery timepoints. Evaluation of donor and recipient microbiota will be by performed by 16S rRNA gene sequencing methodologies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kidney transplant live-donor: Participants that will be a planned live renal transplant donor
  Interventions: Other: Pre-operative assessment - blood, urine, & faecal sample; Other: Post-operative day 3 assessment - blood, urine, & faecal sample; Other: Post-operative week 4-6 assessment - blood, urine, & faecal sample; Other: Post-operative 3 month assessment - blood, urine, & faecal sample; Other: Pre-operative 6 month assessment - blood, urine, & faecal sample; Other: Post-operative month 12 recipient assessment - blood, urine, & faecal sample
- Kidney transplant recipient: Renal transplant recipient on the waiting list to have or will have had an ABO-blood group compatible live-donor or cadaveric transplant
  Interventions: Other: Pre-operative assessment - blood, urine, & faecal sample; Other: Post-operative week 4-6 assessment - blood, urine, & faecal sample; Other: Post-operative 3 month assessment - blood, urine, & faecal sample; Other: Pre-operative 6 month assessment - blood, urine, & faecal sample; Other: Post-operative month 12 recipient assessment - blood, urine, & faecal sample

INTERVENTIONS:
Other: Pre-operative assessment - blood, urine, & faecal sample — Blood sample for multi-parametric flow cytometry. Blood and urine samples for identifying microbial-associated metabolite signature.
  Urine and faecal samples for 16S rRNA gene sequencing
Other: Post-operative day 3 assessment - blood, urine, & faecal sample — Blood sample for multi-parametric flow cytometry. Blood and urine samples for identifying microbial-associated metabolite signature.
  Urine and faecal samples for 16S rRNA gene sequencing.
  Groups: Kidney transplant live-donor
Other: Post-operative week 4-6 assessment - blood, urine, & faecal sample — Blood sample for multi-parametric flow cytometry. Blood and urine samples for identifying microbial-associated metabolite signature.
  Urine and faecal samples for 16S rRNA gene sequencing.
Other: Post-operative 3 month assessment - blood, urine, & faecal sample — Blood sample for multi-parametric flow cytometry. Blood and urine samples for identifying microbial-associated metabolite signature.
  Urine and faecal samples for 16S rRNA gene sequencing.
Other: Pre-operative 6 month assessment - blood, urine, & faecal sample — Blood sample for multi-parametric flow cytometry. Blood and urine samples for identifying microbial-associated metabolite signature.
  Urine and faecal samples for 16S rRNA gene sequencing.
Other: Post-operative month 12 recipient assessment - blood, urine, & faecal sample — Blood sample for multi-parametric flow cytometry. Blood and urine samples for identifying microbial-associated metabolite signature.
  Urine and faecal samples for 16S rRNA gene sequencing.

SUMMARY:
The human gastrointestinal tract harbours ~40 trillion microbial cells, far outnumbering the cell number, and therefore the genetic content of its host. How this genetically diverse bacterial (collectively referred as 'microbiota') co-resident modulates host homeostasis is largely unknown. We are increasing gaining a better understanding how the microbes modulate mucosal and systemic metabolic/immune and organ systems including the kidney, heart and the brain. Therapeutic targeting of the gastrointestinal (GI) microbiota may help improve clinical outcomes in conditions as diverse as arthritis, cardiovascular disease, and cancer. In contrast to other organ systems, studies investigating the role of the microbiota in modulating clinical outcomes in renal transplantation lags behind.

The aim of the study is to examine (a) how alterations in the urinary and GI microbiota and associated metabolites impact on host immunity after renal transplantation, and (b) whether such changes are correlated with post-transplant complications, such as rejection, development of de novo donor specific antibodies, metabolic complications (e.g post-transplant diabetes) and infections. Participants will be followed before and up to twelve months post-transplantation, and, longitudinal microbial data will be correlated with in-depth immune phenotyping and clinical end-points to define the impact that changes in urinary and GI microbial ecology have on kidney transplant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* All adult (≥18 years old) undergoing living donor nephrectomy or kidney transplantation. Patients willing to provide samples including Urine, Blood, Faecal samples.

  1. Participant able to give Informed Consent
  2. All patients will be at least 18 years old
  3. Patients will either be a live renal transplant donor or a renal transplant recipient on the waiting list to have or will have had an ABO-blood group compatible renal transplant.
  4. Patients attending hospital clinics at participating centre for routine clinical follow -up.
  5. Patients willing to comply with study procedures and willing to provide blood, faecal and urine samples.

Exclusion Criteria:

1. Patients under the age of 18 years
2. Patients unable to give informed consent
3. Patients not able to comply with study procedures or follow-up visits
4. Patients that are not a live renal donor or that are not on the waiting list to have or have not had an ABO blood group compatible renal transplant and are not attending hospital outpatient clinics at participating study centres for routine clinical follow-up.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Renal transplant live-donors and recipients of live-donor and cadaveric renal transplants
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in gastrointestinal and urinary microbiota composition and diversity | 1 year
  To understand the overall impact of transplantation on changes to the urinary and GI microbiota, the relative abundance of bacterial taxa will be evaluated using 16S rRNA gene sequencing methodologies. Alpha and Beta diversity indices will be determined from urine samples and faecal samples before and after live-donation and transplantation.
Correlation of change in gastrointestinal and urinary microbiota diversity with post-transplantation outcomes. | 1 year
  Incidence of renal graft dysfunction will be determined by the Modification of Diet in Renal Disease (MDRD)-derived estimated Glomerular Filtration Rate (eGFR) at 12 months.
  Graft survival time - date of transplantation to date of irreversible graft failure signified by return to dialysis (or re-transplantation, whichever is earlier) or the date of last follow-up during the period when the transplant was still functioning. In the event of death with a functioning graft, the follow-up period will be censored at the date of death.

SECONDARY OUTCOMES:
Change in frequency of conventional and regulatory immune phenotypes and correlation with clinical outcome and microbial diversity changes | 1 year
  A panel of validated immune monitoring assays (including multi-colour flow cytometry, intracellular cytokine staining, enzyme-linked immune absorbent spot [ELISpot], enzyme-linked immunosorbent assay [ELISA] and transcriptional analysis) will be used to analyse immunological parameters in patient samples.
Change in microbial-associated metabolite profile and correlation with clinical outcomes and/or microbial diversity changes | 1 year
  A combination of 1H nuclear magnetic resonance (NMR) spectroscopy and liquid chromatography-mass spectrometry will be used to measure the metabolic phenotype of urine and faecal samples from transplant donors and recipients (pre-operatively and up to 12 months after surgery).
Incidence of renal graft dysfunction as determined by the MDRD-derived estimated Glomerular Filtration Rate (eGFR). | 1 year
  A significant deterioration in graft dysfunction is defined as the percent of patients exhibiting an eGFR <45 mL/min/1.73m2 at month 12 or a decrease in eGFR ≥10 mL/min/1.73m2 from month 3 to month 12 after transplantation.
The proportion of patients reaching a defined CKD stage at up to 5 years after transplantation. | 5 years
  Defined by the kidney disease outcomes quality initiative for CKD stages, with eGFR <30 mL/min/1.73m2 considered to be advanced renal dysfunction.
Incidence of biopsy proven acute or chronic cellular or humoral rejection up to 5 years after transplantation as per Banff classification | 5 years
  Revised Banff 2017 classification of antibody-mediated rejection and T cell-mediated rejection in renal allografts.
Incidence of post-donation and post-transplant bacterial or viral infections up to 5 years after surgery | 5 years
  Infectious complications will include, but not be limited to, urinary tract infections (defined as a positive urine culture [>50,000 CFUs/ml] from mid-stream urine, and categorised as asymptomatic bacteriuria [no symptoms], cystitis [lower urinary tract symptoms without systemic features] or pyelonephritis [systemic features, graft dysfunction, CRP>50]), BK viraemia, cytomegalovirus (CMV) viraemia, and respiratory tract (RV) infections.
Patient and graft survival rates up to 5 years after transplantation. | 5 years
  Graft survival time will be calculated from the date of transplantation to the date of irreversible graft failure signified by return to dialysis (or re-transplantation, whichever is earlier) or the date of last follow-up during the period when the transplant was still functioning. In the event of death with a functioning graft, the follow-up period will be censored at the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Research and Development Manager, Study Chair — Sponsor GmbH
Locations (1):
- Royal Free London NHS Trust, London, United Kingdom

DOCUMENTS (1):
  • Informed Consent Form (2020-01-08): https://cdn.clinicaltrials.gov/large-docs/30/NCT04388930/ICF_000.pdf